CLINICAL TRIAL: NCT05820256
Title: Investigating the Effects of Milk Protein Versus Soy Protein on Essential Omega-3 Fatty Acid Metabolism: A Randomized Parallel-arm Human Trial in Healthy Canadian Adults
Brief Title: The Effects of Milk Protein Versus Soy Protein on Essential Omega-3 Fatty Acid Metabolism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, David M Mutch, Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Dietary Proteins and Omega-3s
Record Dates: First submitted 2023-04-03; First posted 2023-04-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Nutrition, Healthy
Keywords: omega-3 metabolism; ALA; EPA; DHA; fatty acid desaturase; fat oxidation
MeSH Terms: interventions — Soybean Proteins

STUDY DESIGN:
Intervention Model Description: Study participants will be block randomized by gender into one of two groups for a parallel-arm trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk Protein Isolate (MPI) (Experimental): Study participants in the MPI group will consume 2 smoothies per day for 31 days, where each smoothie provides 300 kcal in total, composed of 45% from carbohydrate (maltodextrin), 20% from protein (milk protein isolate) and 35% from fat (a blend of flaxseed, safflower, and coconut oils). Each smoothie will be mixed with water up to volume of 250mL. Individuals in this group will not consume soy-containing beverages and foods during the 31-day study.
  Interventions: Dietary Supplement: Milk Protein Isolate (MPI)
- Soy Protein Isolate (SPI) (Experimental): Study participants in the SPI group will consume 2 smoothies per day for 31 days, where each smoothie provides 300 kcal in total, composed of 45% from carbohydrate (maltodextrin), 20% from protein (soy protein isolate) and 35% from fat (a blend of flaxseed, safflower, and coconut oils). Each smoothie will be mixed with water up to volume of 250mL. Individuals in this group will not consume dairy-containing beverages and foods during the 31-day study.
  Interventions: Dietary Supplement: Soy Protein Isolate (SPI)

INTERVENTIONS:
Dietary Supplement: Milk Protein Isolate (MPI) — Study participants will consume two smoothies per day containing a milk protein isolate (MPI) for 31 days.
  Arms: Milk Protein Isolate (MPI)
Dietary Supplement: Soy Protein Isolate (SPI) — Study participants will consume two smoothies per day containing a soy protein isolate (SPI) for 31 days.
  Arms: Soy Protein Isolate (SPI)

SUMMARY:
Dairy products provide macronutrients, vitamins, and minerals that are important for health and development. Despite this, many Canadians now eat fewer dairy products and are instead consuming more non-dairy alternatives, such as soy. Some of this is because of misconceptions about the effects of dairy on health. However, the study investigators hypothesize that, compared to soy, dairy may actually improve a person's health due to its effects on the enzymes in the body that make omega-3 fatty acids, such as EPA and DHA. The goal of this study is to examine omega-3 metabolism in men and women consuming either milk or soy protein. Briefly, this study will determine if the consumption of milk or soy protein differentially impacts blood EPA and DHA levels, the synthesis of EPA and DHA, fatty acid oxidation, and omega-3 fat absorption from the gut. It is anticipated that the findings from this novel and innovative research project will provide high quality evidence to support a previously unappreciated protective effect of dairy for human health and development.

DETAILED DESCRIPTION:
Direct comparisons between dairy and non-dairy plant-based alternatives on metabolic processes in humans are limiting. The study investigators recently completed a cross-sectional analysis in over 1000 young Canadian adult men and women and reported that the consumption of soy beverages/foods was associated with a reduction in estimated fatty acid desaturase pathway activity compared to milk and dairy food consumption (PMID: 34444977). The fatty acid desaturase pathway controls the endogenous synthesis of beneficial long-chain omega-3 polyunsaturated fatty acids (n3-LCPUFA), such as eicosapentaenoic and docosahexaenoic acids (EPA and DHA), from the essential fatty acid, alpha-linolenic acid (ALA). Epidemiological and clinical studies have reported that higher levels of EPA and DHA in the body are associated with reduced CVD risk. Thus, this prior work identified a previously unrecognized cardio-protective role for dairy that could help to counter consumer misconceptions about dairy increasing cardiovascular disease (CVD) risk.

The primary outcome of this research proposal is to determine if the consumption of dairy protein supports n3-LCPUFA synthesis compared to soy protein. The investigators hypothesize that study participants consuming dairy protein will show a greater conversion of ALA into EPA and DHA via the fatty acid desaturase pathway compared to study participants consuming soy protein. To test this hypothesis, the investigators will conduct a randomized, parallel-arm clinical trial in healthy adult men and women who are consuming either a diet containing milk protein isolate (and no soy) or a diet containing soy protein isolate (and no dairy).

Additional secondary outcomes of interest to further advance understanding of how milk and soy proteins affect acute and chronic ALA metabolism will include:

1. Whole blood gene expression analysis of fatty acid desaturases and elongases to determine if milk and soy proteins influence n3-LCPUFA synthesis through a transcriptional mechanism.
2. Breath sample analysis to determine if milk and soy proteins influence ALA degradation through β-oxidation.
3. An oral fat tolerance test (OFTT) to examine if milk and soy proteins modify ALA absorption from the gut.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and pre-menopausal women
* Must be able to consume soy and dairy beverages and foods
* Sufficient level of education to understand study procedures and be able to communicate with clinical staff

Exclusion Criteria:

* Diabetic
* Body mass index greater than 35 kg/m2
* Pregnant or lactating
* Neuropsychiatric disorders (major depression, schizophrenia)
* Digestive disorders
* Inflammatory disease
* Cardiovascular disease
* Use of omega-3 supplements within the last 3 months
* Regular consumption of oily fish
* Allergies/sensitivities to dairy and/or soy food products
* Use of lipid-lowering or digestive medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma EPA and DHA content from baseline | Measured on days: 0 (baseline), 15, 17, 19, 22, 24, 26, 29, 30, and 31
  The change in plasma EPA and DHA content from baseline will be determined by using gas chromatography at multiple time points during the 31-day dietary intervention in which study participants consume 2 smoothies per day containing either a milk protein isolate (MPI) or a soy protein isolate (SPI).

SECONDARY OUTCOMES:
Change in EPA and DHA synthesis from baseline | Measured on days: 0 (baseline), 15, 17, 19, 22, 24, 26, 29, 30, and 31
  The 13-C isotopic signature of EPA and DHA will be measured at Day 0 (baseline) using isotope ratio mass spectrometry (IRMS) to determine a baseline signature. After this baseline measurement, study participants will consume 2 smoothies per day for 31 days containing either SPI or MPI. From days 15 to 31, the smoothies will contain a small amount of an ALA tracer with a defined 13-C isotopic signature. The change in EPA and DHA isotopic signatures will be analyzed at multiple time points during the 31-day intervention by IRMS.
Change in whole blood gene expression from baseline | Measured on days: 0 (baseline) and 31
  Total RNA will be isolated from fasted whole blood samples collected before and after the 31-day dietary intervention from all study participants using a commercially available kit. Total RNA will be used to measure the change in expression of fatty acid desaturase and elongase genes (from baseline) by reverse transcriptase quantitative real time PCR (RT-qPCR).
Change in fatty acid oxidation from baseline | Measured on days: 0 (baseline), 15, 30, and 31
  The 13-C levels in breath samples will be measured at several time point during the dietary intervention to determine the change in ALA oxidation. Basal levels of 13-C in the breath will be determined at Days 0 (baseline) and 15. Starting at Day 15, the daily smoothies consumed by study participants will contain a small amount of an ALA tracer with a defined 13-C isotopic signature. At the end of the intervention, 13-C levels in breath samples will be measured to determine if either the MPI or SPI altered ALA beta-oxidation.
Change in ALA absorption from balance | Measured on days: 0 (baseline) and 31
  An oral fat tolerance test (OFTT) will be used to examine if milk and soy proteins change ALA absorption from the gut. The OFTT will be conducted on Days 0 (baseline) and 31 (end of study). Briefly, study participants will consume a standardized liquid emulsion meal containing 50 g fat (from flaxseed oil, which is rich in plant-based omega-3) and either MPI or SPI. Study participants will consume this liquid meal within 15 minutes. Blood samples will be collected hourly during the OFTT and ALA content in the chylomicron rich fraction will be measured by gas chromatography.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Guelph, Guelph, Ontario
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be anonymized.

REFERENCES:
- [Background] Gonzalez-Soto M, Abdelmagid SA, Ma DWL, El-Sohemy A, Mutch DM. Soy Consumption, but Not Dairy Consumption, Is Inversely Associated with Fatty Acid Desaturase Activity in Young Adults. Nutrients. 2021 Aug 17;13(8):2817. doi: 10.3390/nu13082817. PMID 34444977